CLINICAL TRIAL: NCT01459640
Title: Phase 2 Study Assessing the Efficacy of Intra-Articular Autologous Mesenchymal Stem Cells in Patients With Mild to Moderate Osteoarthritis
Brief Title: Intra-Articular Autologous Bone Marrow Mesenchymal Stem Cells Transplantation to Treat Mild to Moderate Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Cytopeutics Pte. Ltd. (Industry)
Responsible Party: Principal Investigator, Dr Ya Mohammad Hassan Shukur, Senior Consultant Orthopedic Surgeon, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FF-114-2011
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Bone marrow; Mesenchymal stem cells; Autologous; Mild osteoarthritis; Moderate osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid; orthovisc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronic acid (Active Comparator)
  Interventions: Drug: Hyaluronic Acid
- Bone marrow mesenchymal stem cells (Experimental): Autologous bone marrow-derived mesenchymal stem cells
  Interventions: Biological: Autologous bone marrow-derived mesenchymal stem cells

INTERVENTIONS:
Drug: Hyaluronic Acid — Intra-articular injection; 30mg/2ml; three-weekly injection regimen
  Other Names: Orthovisc
  Arms: Hyaluronic acid
Biological: Autologous bone marrow-derived mesenchymal stem cells — Single intra-articular implantation of autologous bone marrow-derived mesenchymal stem cells in hyaluronic acid "Orthovisc" (3rd injection in a three-weekly injection regimen)
  Arms: Bone marrow mesenchymal stem cells

SUMMARY:
Osteoarthritis is a progressively degenerative disease resulting in increasing pain, impairment and ultimately disability. While the available treatments seek to ameliorate pain or improve mobility, these treatments rarely modify the course of the disease, but rather attend to its consequences. For early stage osteoarthritis, treatment is largely limited to addressing the symptoms of inflammation with non-steroidal anti-inflammatory drugs (NSAIDs). These drugs do not stop the progression of the condition or regenerates damaged cartilage.

This is a randomized and open labelled study aimed to determine the efficacy of intra-articular implantation of autologous bone marrow-derived mesenchymal stem cells in patients with mild to moderate osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild to moderate osteoarthritis based on Kellgren-Lawrence radiographic classification
* Has a history of joint swelling, pain, stiffness, altered gait and loss of motion due to degenerative cartilage

Exclusion Criteria:

* Has systemic bone or cartilage disorders
* Has significant vascular impairment proximal to implant site
* Has substantial joint destabilization including extensive osteophyte formation
* Has substantial surface erosion of the weight-bearing articular cartilage
* Evidence of infection or fractures in or around the joint
* Contraindication to bone marrow aspiration
* Any acute or chronic communicable diseases including Hepatitis B, Hepatitis C and HIV
* Any past history of neoplasia and primary hematological disease
* Renal impairment indicated by serum creatinine greater than 200mM
* Liver impairment indicated by serum aspartate transaminase and serum alanine transaminase greater than 120 IU
* Any other co-morbidity which the physician deems as a contraindication to stem cell transplantation and bone marrow biopsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cartilage thickness at 12 months by MRI | 12 months

SECONDARY OUTCOMES:
Visual Analog Score | 1 month, 3 months, 6 months, 9 months, 12 months
IKDC Subjective Knee Evaluation Form (2000) | 1 month, 3 months, 6 months, 9 months, 12 months
Change from baseline in progression of osteoarthritis at 12 months by plain radiograph (X-ray) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ya Mohammad Hassan Shukur, MD, Principal Investigator — UKM Medical Centre
Locations (1):
- UKM Medical Centre, Kuala Lumpur, Malaysia